CLINICAL TRIAL: NCT02736942
Title: COLOR III: A Multicentre Randomised Clinical Trial Comparing Transanal TME Versus Laparoscopic TME for Mid and Low Rectal Cancer
Brief Title: COLOR III Trial: Transanal vs Laparoscopic TME
Acronym: COLORIII
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, H.J. Bonjer, Professor of Surgery, MD, PhD, FRCSC, Amsterdam UMC, location VUmc
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015.449
Record Dates: First submitted 2016-02-18; First posted 2016-04-13 (Estimated); Last update posted 2019-06-06 (Actual); Status verified 2019-06

CONDITIONS: Rectal Carcinoma; Surgery
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Laparoscopic (Active Comparator): Laparoscopic TME
  Interventions: Procedure: Laparoscopic TME
- Transanal (Experimental): TaTME
  Interventions: Procedure: TaTME

INTERVENTIONS:
Procedure: Laparoscopic TME — Laparoscopic Total Mesorectal Excision
  Arms: Laparoscopic
Procedure: TaTME — Transanal Total Mesorectal Excision
  Arms: Transanal

SUMMARY:
Background Surgery for mid and low rectal cancer is associated with relative high rates of incomplete mesorectal excisions and high rates of circumferential resection margin (CRM) involvement resulting in significant number of local recurrences. Moreover, patients with mid and low rectal cancer suffer from high rates of morbidity, permanent colostomies and impairment of quality of life. The transanal TME (TaTME) has been developed to improve the quality of TME surgery in mid and low rectal cancer.

Study design The COLOR III trial is an international multicentre randomised study comparing short- and long-term outcomes of TaTME and laparoscopic TME for rectal cancer. The study will include a quality assessment phase before randomisation to ensure required competency level and uniformity of the new TaTME technique and the laparoscopic TME. During the trial clinical data will be reviewed centrally to ensure uniform quality.

Endpoints The primary endpoint of the study is the local recurrence rate at 3-years follow-up. Secondary endpoints include sphincter saving procedures, short-term morbidity and mortality, involved circumferential resection margin (CRM), disease-free and overall survival at 3 and 5 years, completeness of mesorectum and quality of life.

Statistics In laparoscopic TME the percentage of local recurrence at 3-years follow-up is estimated 5%. With the non-inferiority margin set at 4%, with a one-sided level of significance of 2.5% and a power of 80%, a total of 1104 patients is needed, 669 patients in the TaTME arm and 335 patients in the laparoscopic TME arm. All analyses will be performed on intention-to-treat basis.

Main selection criteria Patients with histologically proven single mid or distal rectum carcinoma (0 to 10 cm from anal verge) at MRI, eligible for restorative surgery with a curative intent, are included. Patients with a T1 tumor suitable for local excision, T3 tumors with a suspected involved circumferential resection margin and T4 tumors are excluded.

Hypothesis The hypothesis is that TaTME will result in a comparable local recurrence rate at 3-years follow-up with benefit of lower morbidity and conversions. Furthermore, because of direct endoscopic visualization, even in very low tumors a coloanal anastomosis can be created, resulting in a lower colostomy rate compared with laparoscopic and open resection. Because long-term outcomes are unknown, within a trial setting the technique can be standardized and quality control can be performed.

DETAILED DESCRIPTION:
To improve oncological and functional outcomes of patients with rectal cancer new surgical techniques are being developed. The adoption of the TME technique has resulted in better oncological outcome in the last decades. The addition of neoadjuvant therapy has further improved oncological outcome. The minimal invasive laparoscopic resection of rectal cancer has shown to be safe and to result in improved short-term outcomes and reduced morbidity.

Nevertheless, the laparoscopic resection of mid and low rectal cancer remains challenging due to the anatomy of the narrow pelvis and is associated with a relative high risk of resections with an involved CRM resulting in increased risk of a local recurrence.

In attempt to improve the quality of the TME procedure in low rectal cancer and further improve oncological results the TaTME has been developed, in which the rectum is dissected transanally according to TME principles. First series have been described since 2010 and although randomised evidence is still lacking this new technique has shown to be feasible and safe. The rectum including the total mesorectum is mobilised transanally in a reversed way with minimally invasive surgery including high quality imaging techniques.

The TaTME technique for mid and low rectal cancer has shown to have potential benefits: better specimen quality with less R1 resections, less morbidity, less conversion to laparotomy and more sphincter saving rectal resections without compromising oncological outcomes.

The investigators propose to evaluate the TaTME technique compared with conventional laparoscopic rectal resection for patients with mid and low rectal cancer in an international randomised trial: the COLOR III trial.

ELIGIBILITY:
Inclusion Criteria:

* Solitary mid (5.1-10cm from anal verge on MRI) or low (0-5cm from anal verge on MRI) rectal cancer observed at colonoscopy and histologically proven through biopsy
* Distal border of the tumour within 10cm from the anal verge on MRI-scan
* Tumour with threatened margins downstaged after neoadjuvant therapy to free margins
* No evidence for distal metastases on imaging of thorax and abdomen
* Suitable for elective surgical resection
* Informed consent according to local requirements

Exclusion Criteria:

* T3 tumours with margins less than 1mm to the MRF, determined by MRI-scan (as staged after preoperative chemo- and/or radiotherapy)
* T4 tumours, as staged after preoperative chemo- and/or radiotherapy
* Tumours with in growth more than 1/3 of anal sphincter complex or levator ani
* Malignancy other than adenocarcinoma at histological examination
* Patients under 18 years of age
* Pregnancy
* Previous rectal surgery (excluding local excision, EMR (endoscopic mucosal resection) or polypectomy)
* Signs of acute intestinal obstruction
* Multiple colorectal tumours
* Familial Adenomatosis Polyposis Coli (FAP), Hereditary Non-Polyposis Colorectal Cancer (HNPCC), active Crohn's disease or active ulcerative colitis
* Planned synchronous abdominal organ resections
* Preoperative suspicion of invasion of adjacent organs through MRI-scan
* Preoperative evidence for distant metastases through imaging of the thorax and abdomen
* Other malignancies in medical history, except adequately treated basocellular carcinoma of the skin or in situ carcinoma of the cervix uteri
* Absolute contraindications to general anaesthesia or prolonged pneumoperitoneum, as severe cardiovascular or respiratory disease (ASA class > III)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1104 (Estimated)
Dates: Start 2016-12-02 (Actual); Primary Completion 2021-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Local recurrence rate | 3 years
  Local recurrence rate, determined by MRI at 3 year follow-up

SECONDARY OUTCOMES:
Percentage of participants with involvement of circumferential resection margin (tumour cells < 1mm from circumferential resection margin) | Post operative 1 month
  Pathological microscopic examination of specimen
Morbidity rate | 5 years
Mortality rate | 5 years
Percentage of participants with recurrence | 5 years
  Local and distant.
Disease-free survival rate | 5 years
Overall survival rate | 5 years
Percentage of sphincter saving procedures | 4 years
Change in functional outcomes (LARS questionnaire) | Baseline and 1 year
  Measured by questionnaires
Change in Health Related Quality of Life (EORTC QLQ-29 questionnaire) | Baseline and 1 year
  Measured by questionnaires
Change in Health Related Quality of Life (EORTC QLQ-30 questionnaire) | Baseline and 1 year
  Measured by questionnaires
Change in Health Related Quality of Life (EQ 5-D questionnaire) | Baseline and 1 year
  Measured by questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Hendrik J. Bonjer, MD, PhD, Principal Investigator — Amsterdam UMC, location VUmc; Antonio M. Lacy, MD, PhD, Principal Investigator — Hospital Clinic of Barcelona; George B. Hanna, MD, PhD, Principal Investigator — Imperial College London; Jurriaan B. Tuynman, MD, PhD, Study Director — Amsterdam UMC, location VUmc; Colin Sietses, MD, PhD, Study Director — Gelderse Vallei Hospital Ede
Locations (1):
- VU University Medical Center, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No
We are not sharing confidential individual patient data.

REFERENCES:
- See also: Official trial website — http://www.color3trial.com